CLINICAL TRIAL: NCT01575769
Title: Long-term, Interventional, Open Label Extension Study Evaluating the Safety of Tocilizumab Treatment in Patients With Polyarticular-course Juvenile Idiopathic Arthritis From Poland and Russia Who Completed the Global, Multinational Trial (WA19977).
Brief Title: An Extension Study to WA19977 in Patients With Active Polyarticular-Course Juvenile Idiopathic Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prior to the planned final on-treatment efficacy assessments due to commercial availability of tocilizumab in Russia and Poland.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML27783
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2017-08

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RoActemra/Actemra (tocilizumab)

INTERVENTIONS:
Drug: RoActemra/Actemra (tocilizumab) — Tocilizumab 8 mg/kg every 4 weeks for 104 weeks

SUMMARY:
This long-term, interventional, open-label extension study will evaluate the safety and efficacy of RoActemra/Actemra (tocilizumab) in patients from Poland and Russia with polyarticular-course juvenile idiopathic arthritis who completed the WA19977 study. Patients will receive RoActemra/Actemra 8 mg/kg every 4 weeks. The anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed 104 weeks of study WA19977 with at least a JIA ACR30 clinical response to RoActemra/Actemra and no serious adverse event or adverse event
* Written informed consent obtained from patient if patient is 18 years of age and older, or if under the age of 18 years from parents or legal guardian

Exclusion Criteria:

* Patient did not benefit from RoActemra/Actemra therapy in study WA19977
* Treatment with any investigational drug since the last administration of study drug in the core study WA19977
* Patients developed any other autoimmune rheumatic disease other than the permitted JIA subsets
* Any significant medical or surgical condition that would jeopardize patient's safety
* Current serious uncontrolled concomitant disease or infection

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-01-19 (Actual); Primary Completion 2013-12-03 (Actual); Study Completion 2013-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Poland (5):
  - Wojewodzki Szpital Dzieciecy Im. J. Brudzinskiego, Bydgoszcz
  - Wojewodzki Specjalistyczny Szpital Dzieciecy Sw Ludwika; Oddzial Dzieci Starszych, Krakow
  - Uniwersytecki Szpital Kliniczny Nr 4 im. M. Konopnickiej; Oddz. Kardiolog. i Reumatolog. dla Dzieci, Lodz
  - Dzieciecy Szpital Kliniczny IM. Prof. A. Gebali; Oddzial Pediatrii Chorob Pluc I Reumatologii, Lublin
  - Centrum Pediatrii im Jana Pawla II; Oddzial Reumatologiczny, Sosnowiec
- Russia (6):
  - Scientific Research Institute, Moscow
  - SBEI of HPI The 1st Moscow State Medical University n.a. I.M. Sechenov of MOH of RF, Moscow
  - SI Sceintific children health center RAMS, Moscow
  - GOU VPO Rostovskiy state medical university Roszdrav, Rostov-on-Don
  - Saint-Petersburg State; Pediatrics Medical Academy, Saint Petersburg
  - Samara Regional Clinical Cardiology Dispensary, Samara

REFERENCES:
- [Derived] Opoka-Winiarska V, Zuber Z, Alexeeva E, Chasnyk V, Nikishina I, Debowska G, Smolewska E. Long-term, interventional, open-label extension study evaluating the safety of tocilizumab treatment in patients with polyarticular-course juvenile idiopathic arthritis from Poland and Russia who completed the global, international CHERISH trial. Clin Rheumatol. 2018 Jul;37(7):1807-1816. doi: 10.1007/s10067-018-4071-9. Epub 2018 Apr 13. PMID 29654485

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed Visit 33 (Week 104) of the core study WA19977 (NCT00988221) with at least juvenile idiopathic arthritis (JIA) American College of Rheumatology (ACR) 30 clinical response were eligible to continue the study therapy within this long-term extension study in Russia and Poland.
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilograms (mg/kg) via intravenous (IV) infusion, once every 4 weeks for up to 104 weeks or until tocilizumab became commercially available, whichever occurred first.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 41
Completed | 0
Not Completed | 41
Not completed — Adverse Event | 1
Not completed — Study terminated by sponsor | 40

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who entered the study, took at least one dose of study drug, and with at least one safety follow-up, regardless of premature withdrawal.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg via IV infusion, once every 4 weeks for up to 104 weeks or until tocilizumab became commercially available, whichever occurred first.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: AE: unfavorable and unintended sign, symptom, or disease associated with use of treatment, regardless of treatment relation. Pre-existing conditions that worsened and laboratory or clinical tests that resulted in change in treatment or discontinuation from treatment were reported as AEs. Serious AE: resulted in death, life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect or was medically significant. Severe AE: AE that caused inability to work or perform normal daily activity. AEs of special interest: Serious infections (including opportunistic infections), Myocardial infarction/Acute coronary syndrome, Gastrointestinal perforations and related AE, Malignant neoplasms, Anaphylaxis event, Demyelination-related events, Stroke, Spontaneous or serious bleeding, Serious/medically significant hepatic events. Any AE included serious and non-serious AE.
Time Frame: Baseline to 12 weeks after last actual study medication (up to 101 weeks)
Population: Safety population
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg via IV infusion,once every 4 weeks for up to 104 weeks or until tocilizumab became commercially available, whichever occurred first.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Any AEs | 56.1
  Any Treatment Related AEs | 29.3
  Any SAEs | 7.3
  Any Severe AEs | 2.4
  Any Life Threatening AEs | 0.0
  AEs of Special Interest | 0.0
  AE Leading to Dosage Modification/Interruption | 22.0
  Withdrawal Due to AEs | 2.4
  Withdrawal Due to SAEs | 2.4
  Withdrawal Due to AEs of Special Interest | 0.0

2. Secondary Outcome: Percentage of Participants With JIA ACR 30 Response at Weeks 12, 24 and End of Follow Up
Description: JIA ACR30 response was defined as 3 of any 6 core outcome variables improved by at least 30% of the baseline assessments, with no more than 1 of the remaining variables worsened by more than 30%. Six core variables were: Physician global assessment (PGA) of disease activity using Visual Analog Scale (VAS) from left end of line 0 (inactive arthritis) to right end of line 100 (very active arthritis); Patient/parent global assessment (PtGA) of overall well-being using a VAS from left end of line 0 (very well) to right end of line 100 (very poor); Number of joints with active arthritis (joints with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both); Number of joints with limitation of movement; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and Erythrocyte Sedimentation Rate (ESR).
Time Frame: Baseline, Week 12, 24, End of Follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg via IV infusion, once every 4 weeks for up to 104 weeks or until tocilizumab became commercially available whichever, occurred first.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Baseline | 100.0 [91.4 to 100.0]
  Week 12 | 100.0 [91.4 to 100.0]
  Week 24 | 100.0 [91.4 to 100.0]
  Follow up | 80.5 [65.1 to 91.2]

3. Secondary Outcome: Percentage of Participants With JIA ACR 50 Response at Weeks 12, 24 and End of Follow up
Description: JIA ACR50 response was defined as 3 of any 6 core outcome variables improved by at least 50% of the baseline assessments, with no more than 1 of the remaining variables worsened by more than 30%. Six core variables were: PGA of disease activity using VAS from left end of line 0 (inactive arthritis) to right end of line 100 (very active arthritis); PtGA of overall well-being using a VAS from left end of line 0 (very well) to right end of line 100 (very poor); Number of joints with active arthritis (joints with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both); Number of joints with limitation of movement; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and ESR.
Time Frame: Baseline, Week 12, 24, End of Follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Baseline | 100.0 [91.4 to 100.0]
  Week 12 | 100.0 [91.4 to 100.0]
  Week 24 | 100.0 [91.4 to 100.0]
  Follow up | 80.5 [65.1 to 91.2]

4. Secondary Outcome: Percentage of Participants With JIA ACR 70 Response at Weeks 12, 24 and End of Follow up
Description: JIA ACR70 response was defined as 3 of any 6 core outcome variables improved by at least 70% of the baseline assessments, with no more than 1 of the remaining variables worsened by more than 30%. Six core variables were: PGA of disease activity using VAS from left end of line 0 (inactive arthritis) to right end of line 100 (very active arthritis); PtGA of overall well-being using a VAS from left end of line 0 (very well) to right end of line 100 (very poor); Number of joints with active arthritis (joints with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both); Number of joints with limitation of movement; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and ESR
Time Frame: Baseline, Week 12, 24, End of Follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Baseline | 100.0 [91.4 to 100.0]
  Week 12 | 100.0 [91.4 to 100.0]
  Week 24 | 97.6 [87.1 to 99.9]
  Follow up | 78.0 [62.4 to 89.4]

5. Secondary Outcome: Percentage of Participants With JIA ACR 90 Response at Weeks 12, 24 and End of Follow up
Description: JIA ACR90 response was defined as 3 of any 6 core outcome variables improved by at least 90% of the baseline assessments, with no more than 1 of the remaining variables worsened by more than 30%. Six core variables were: PGA of disease activity using VAS from left end of line 0 (inactive arthritis) to right end of line 100 (very active arthritis); PtGA of overall well-being using a VAS from left end of line 0 (very well) to right end of line 100 (very poor); Number of joints with active arthritis (joints with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both); Number of joints with limitation of movement; Health Assessment Questionnaire: 20 questions in 8 areas (dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities) answered on a scale of 0=without difficulty to 3=unable to do; and ESR.
Time Frame: Baseline, Week 12, 24, End of Follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Baseline | 73.2 [57.1 to 85.8]
  Week 12 | 78.0 [62.4 to 89.4]
  Week 24 | 80.5 [65.1 to 91.2]
  Follow up | 75.6 [59.7 to 87.6]

6. Secondary Outcome: Percentage of Participants With Inactive Disease at Week 12, 24 and End of Follow up
Description: Criteria for Inactive Disease: 1) No joints with active arthritis (joints with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both), 2) No fever, rash, serositis, splenomegaly, hepatomegaly (by physical exam) or generalized lymphadenopathy attributable to systemic juvenile idiopathic arthritis (sJIA), 3) Normal ESR (less than [<] 20 millimeters per hour [mm/hour]), and 4) PGA of disease activity using VAS indicated no disease activity (where no disease activity is considered to be a score less than or equal to [≤]10 mm on a 100 mm VAS where left end of line 0 [inactive arthritis] to right end of line 100 [very active arthritis]).
Time Frame: Baseline, Week 12, 24, End of Follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Baseline | 63.4 [46.9 to 77.9]
  Week 12 | 65.9 [49.4 to 79.9]
  Week 24 | 75.6 [59.7 to 87.6]
  Follow up | 61.0 [44.5 to 75.8]

7. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 12, 24 and End of Follow up
Description: Clinical remission: inactive disease for minimum of 6 continuous months while on medication (Level 1); off oral corticosteroid medications but still on tocilizumab (Level 2); off both methotrexate and oral corticosteroids but still on tocilizumab (Level 3); or off all anti-arthritis medications-oral corticosteroids, methotrexate, non-steroidal anti-inflammatory drugs but still on tocilizumab (Level 4). Inactive disease: No joints with active arthritis (joints with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both); No fever, rash, serositis, splenomegaly, hepatomegaly (by physical exam) or generalized lymphadenopathy attributable to sJIA; Normal ESR (<20 mm/hour); PGA of disease activity indicated no disease activity (score ≤10 mm on a 100 mm VAS where 0 [inactive arthritis] and 100 [very active arthritis]). Overall percentage of participants with clinical remission (any level) are reported.
Time Frame: Baseline, Week 12, 24, End of Follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Baseline | 43.9 [28.5 to 60.3]
  Week 12 | 46.3 [30.7 to 62.6]
  Week 24 | 48.8 [32.9 to 64.9]
  Follow up | 46.3 [30.7 to 62.6]

8. Secondary Outcome: Change From Baseline in Joints With Active Arthritis at Weeks 12, 24, 36, 48, 60, 72, 84, End of Follow up
Description: Joint with active arthritis was defined as a joint with swelling not due to deformity or joints with limitation of motion and with pain, tenderness or both.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
Joints
  Baseline (n=41) | 1.4 (2.68)
  Change From Baseline at Week 12 (n=41) | -0.1 (1.70)
  Change From Baseline at Week 24 (n=41) | -0.4 (4.56)
  Change From Baseline at Week 36 (n=35) | -1.4 (2.80)
  Change From Baseline at Week 48 (n=22) | -1.7 (3.34)
  Change From Baseline at Week 60 (n=17) | 0.4 (8.17)
  Change From Baseline at Week 72 (n=10) | 1.9 (7.52)
  Change From Baseline at Week 84 (n=7) | 3.9 (11.55)
  Change From Baseline at Follow Up (n=33) | 1.2 (4.14)

9. Secondary Outcome: Change From Baseline in Number of Joints With Limitation of Movement at Weeks 12, 24, 36, 48, 60, 72, 84, End of Follow up
Description: The maximum number of joints with limitation of movement is 67 and these were defined as those with 'limitation of motion'.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
Joints
  Baseline (n=41) | 3.5 (6.30)
  Change From Baseline at Week 12 (n=41) | -0.6 (2.23)
  Change From Baseline at Week 24 (n=41) | -0.9 (2.75)
  Change From Baseline at Week 36 (n=35) | -1.3 (3.14)
  Change From Baseline at Week 48 (n=22) | -1.5 (4.21)
  Change From Baseline at Week 60 (n=17) | -1.2 (5.10)
  Change From Baseline at Week 72 (n=10) | 0.0 (1.83)
  Change From Baseline at Week 84 (n=7) | 0.7 (3.09)
  Change From Baseline at Follow Up (n=33) | 2.6 (5.80)

10. Secondary Outcome: Change From Baseline in PGA of Disease Activity at Weeks 12, 24, 36, 48, 60, 72, 84, End of Follow up
Description: The physician provides a rating of the participant's arthritis disease activity on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'arthritis inactive' (ie, symptom-free and no arthritis symptoms) and the extreme right end represents 'arthritis very active'. A higher score indicates more disease activity. A negative change score indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
mm
  Baseline (n=41) | 4.5 (4.99)
  Change From Baseline at Week 12 (n=41) | 1.0 (5.66)
  Change From Baseline at Week 24 (n=41) | 0.1 (4.97)
  Change From Baseline at Week 36 (n=35) | -0.6 (4.29)
  Change From Baseline at Week 48 (n=22) | -0.4 (5.80)
  Change From Baseline at Week 60 (n=17) | 0.4 (6.52)
  Change From Baseline at Week 72 (n=10) | 1.0 (6.50)
  Change From Baseline at Week 84 (n=7) | 2.9 (13.09)
  Change From Baseline at Follow Up (n=33) | 4.4 (8.65)

11. Secondary Outcome: Change From Baseline in PtGA of Overall Well-Being at Weeks 12, 24, 36, 48, 60, 72, 84, End of Follow up
Description: The participant or parent/guardian, as appropriate, provides a rating of the participant's well-being on a 0 to 100 mm horizontal scale. The extreme left end of the line represents 'very well' (ie, symptom-free and no arthritis disease activity) and the extreme right end represents 'very poor' (ie, maximum arthritis disease activity). A higher score indicates poorer well-being. A negative change score indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
mm
  Baseline (n=41) | 4.0 (5.72)
  Change From Baseline at Week 12 (n=41) | -0.2 (3.31)
  Change From Baseline at Week 24 (n=41) | -1.5 (4.38)
  Change From Baseline at Week 36 (n=35) | -2.2 (4.34)
  Change From Baseline at Week 48 (n=22) | -2.2 (4.89)
  Change From Baseline at Week 60 (n=17) | -1.2 (2.08)
  Change From Baseline at Week 72 (n=10) | -0.9 (1.60)
  Change From Baseline at Week 84 (n=7) | -0.9 (2.19)
  Change From Baseline at Follow Up (n=33) | 3.2 (7.39)

12. Secondary Outcome: Change From Baseline in ESR at Weeks 12, 24, 36, 48, 60, 72, 84, End of Follow up
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: millimeters per hour (mm/hour)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
millimeters per hour (mm/hour)
  Baseline (n=41) | 5.0 (4.08)
  Change From Baseline at Week 12 (n=41) | -0.95 (3.83)
  Change From Baseline at Week 24 (n=41) | -0.9 (5.01)
  Change From Baseline at Week 36 (n=35) | -1.2 (5.26)
  Change From Baseline at Week 48 (n=22) | -0.9 (3.30)
  Change From Baseline at Week 60 (n=17) | -0.35 (5.22)
  Change From Baseline at Week 72 (n=10) | 0.5 (6.88)
  Change From Baseline at Week 84 (n=7) | 3.3 (14.68)
  Change From Baseline at Follow Up (n=33) | 5.9 (8.07)

13. Secondary Outcome: Change From Baseline in Childhood Health Assessment - Disability Index (CHAQ-DI) at Weeks 12, 24, 36, 48, 60, 72, 84, End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. To calculate the overall score, the participant must have a domain score in at least 6 of the 8 domains. The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A higher score indicates less ability.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.1 (0.24)
  Change From Baseline at Week 12 (n=41) | -0.0 (0.06)
  Change From Baseline at Week 24 (n=41) | 0.0 (0.09)
  Change From Baseline at Week 36 (n=35) | -0.0 (0.09)
  Change From Baseline at Week 48 (n=22) | -0.1 (0.15)
  Change From Baseline at Week 60 (n=17) | 0.0 (0.08)
  Change From Baseline at Week 72 (n=10) | -0.1 (0.09)
  Change From Baseline at Week 84 (n=7) | -0.1 (0.26)
  Change From Baseline at Follow Up (n=33) | 0.1 (0.25)

14. Secondary Outcome: Percentage of Participants With Minimally Important Improvement in the CHAQ-DI Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. To calculate the overall score, the participant must have a domain score in at least 6 of the 8 domains. The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A higher score indicates less ability. A minimally important improvement was defined as at least a 0.13 improvement in CHAQ-DI score from baseline.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  Week 12 | 2.4 [0.1 to 12.9]
  Week 24 | 2.4 [0.1 to 12.9]
  Week 36 | 5.7 [0.7 to 19.2]
  Week 48 | 18.2 [5.2 to 40.3]
  Week 72 | 10.0 [0.3 to 44.5]
  Week 84 | 28.6 [3.7 to 71.0]
  Follow Up | 15.2 [5.1 to 31.9]

15. Secondary Outcome: Change From Baseline in CHAQ-DI (Activitiy) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Activity component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=40) | 0.2 (0.41)
  Change From Baseline at Week 12 (n=39) | 0.0 (0.16)
  Change From Baseline at Week 24 (n=39) | 0.0 (0.28)
  Change From Baseline at Week 36 (n=34) | 0.0 (0.35)
  Change From Baseline at Week 48 (n=22) | -0.1 (0.35)
  Change From Baseline at Week 60 (n=17) | -0.1 (0.43)
  Change From Baseline at Week 72 (n=10) | -0.1 (0.57)
  Change From Baseline at Week 84 (n=7) | -0.1 (0.38)
  Change From Baseline at Follow Up (n=33) | -0.1 (0.35)

16. Secondary Outcome: Change From Baseline in CHAQ-DI (Arising) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Arising component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.0 (0.22)
  Change From Baseline at Week 12 (n=40) | 0.0 (0.23)
  Change From Baseline at Week 24 (n=40) | 0.0 (0.16)
  Change From Baseline at Week 36 (n=34) | -0.0 (0.17)
  Change From Baseline at Week 48 (n=22) | -0.0 (0.21)
  Change From Baseline at Week 60 (n=17) | -0.1 (0.24)
  Change From Baseline at Week 72 (n=10) | 0.0 (0.0)
  Change From Baseline at Week 84 (n=7) | 0.0 (0.0)
  Change From Baseline at Follow Up (n=33) | 0.0 (0.17)

17. Secondary Outcome: Change From Baseline in CHAQ-DI (Dressing and Grooming) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Dressing and Grooming component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.1 (0.42)
  Change From Baseline at Week 12 (n=40) | 0.0 (0.16)
  Change From Baseline at Week 24 (n=40) | 0.1 (0.22)
  Change From Baseline at Week 36 (n=34) | 0.1 (0.24)
  Change From Baseline at Week 48 (n=22) | 0.0 (0.31)
  Change From Baseline at Week 60 (n=17) | 0.0 (0.35)
  Change From Baseline at Week 72 (n=10) | -0.2 (0.63)
  Change From Baseline at Week 84 (n=7) | -0.3 (0.76)
  Change From Baseline at Follow Up (n=33) | -0.1 (0.50)

18. Secondary Outcome: Change From Baseline in CHAQ-DI (Eating) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Eating component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.1 (0.33)
  Change From Baseline at Week 12 (n=40) | 0.0 (0.23)
  Change From Baseline at Week 24 (n=40) | 0.0 (0.23)
  Change From Baseline at Week 36 (n=34) | 0.0 (0.25)
  Change From Baseline at Week 48 (n=22) | -0.1 (0.29)
  Change From Baseline at Week 60 (n=17) | 0.1 (0.24)
  Change From Baseline at Week 72 (n=10) | 0.0 (0.0)
  Change From Baseline at Week 84 (n=7) | -0.1 (0.38)
  Change From Baseline at Follow Up (n=33) | -0.0 (0.30)

19. Secondary Outcome: Change From Baseline in CHAQ-DI (Grip) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Grip component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.2 (0.40)
  Change From Baseline at Week 12 (n=40) | -0.1 (0.22)
  Change From Baseline at Week 24 (n=40) | -0.0 (0.16)
  Change From Baseline at Week 36 (n=34) | -0.1 (0.29)
  Change From Baseline at Week 48 (n=22) | -0.1 (0.29)
  Change From Baseline at Week 60 (n=17) | 0.1 (0.43)
  Change From Baseline at Week 72 (n=10) | 0.0 (0.47)
  Change From Baseline at Week 84 (n=7) | -0.1 (0.38)
  Change From Baseline at Follow Up (n=33) | -0.1 (0.29)

20. Secondary Outcome: Change From Baseline in CHAQ-DI (Hygiene) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Hygiene component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.2 (0.44)
  Change From Baseline at Week 12 (n=40) | -0.0 (0.16)
  Change From Baseline at Week 24 (n=40) | 0.0 (0.16)
  Change From Baseline at Week 36 (n=34) | -0.1 (0.24)
  Change From Baseline at Week 48 (n=22) | -0.1 (0.35)
  Change From Baseline at Week 60 (n=17) | -0.1 (0.43)
  Change From Baseline at Week 72 (n=10) | -0.1 (0.32)
  Change From Baseline at Week 84 (n=7) | -0.4 (0.79)
  Change From Baseline at Follow Up (n=33) | -0.2 (46)

21. Secondary Outcome: Change From Baseline in CHAQ-DI (Reach) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Reach component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.2 (0.42)
  Change From Baseline at Week 12 (n=40) | -0.0 (0.28)
  Change From Baseline at Week 24 (n=40) | -0.1 (0.22)
  Change From Baseline at Week 36 (n=34) | -0.0 (0.30)
  Change From Baseline at Week 48 (n=22) | -0.1 (0.29)
  Change From Baseline at Week 60 (n=17) | 0.1 (0.43)
  Change From Baseline at Week 72 (n=10) | 0.0 (0.0)
  Change From Baseline at Week 84 (n=7) | 0.0 (0.0)
  Change From Baseline at Follow Up (n=33) | -0.1 (0.38)

22. Secondary Outcome: Change From Baseline in CHAQ-DI (Walking) Score at Weeks 12, 24, 36, 48, 60, 72, 84 and End of Follow up
Description: The CHAQ-DI, as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Walking component was measured on 0-3 scale (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do).
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  Baseline (n=41) | 0.0 (0.16)
  Change From Baseline at Week 12 (n=40) | 0.0 (0.0)
  Change From Baseline at Week 24 (n=40) | 0.1 (0.22)
  Change From Baseline at Week 36 (n=34) | 0.0 (0.0)
  Change From Baseline at Week 48 (n=22) | 0.0 (0.0)
  Change From Baseline at Week 60 (n=17) | 0.1 (0.24)
  Change From Baseline at Week 72 (n=10) | 0.0 (0.0)
  Change From Baseline at Week 84 (n=7) | 0.0 (0.0)
  Change From Baseline at Follow Up (n=33) | 0.0 (0.0)

23. Secondary Outcome: Absolute C-Reactive Protein Levels
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, End of follow up (up to 101 weeks)
Population: Safety population. Here, 'n' signifies the number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: milligrams per Liter
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
milligrams per Liter
  Baseline (n=40) | 0.9468 (4.11395)
  Week 4 (n=39) | 0.9755 (1.71814)
  Week 8 (n=41) | 1.8995 (6.17464)
  Week 12 (n=41) | 1.7157 (3.07714)
  Week 16 (n=41) | 2.4115 (8.71986)
  Week 20 (n=39) | 0.9706 (2.67299)
  Week 24 (n=41) | 1.4893 (3.24038)
  Week 28 (n=40) | 2.2320 (5.51994)
  Week 32 (n=39) | 2.1713 (7.09086)
  Week 36 (n=35) | 1.6507 (4.81621)
  Week 40 (n=31) | 1.2562 (2.49440)
  Week 44 (n=26) | 1.1710 (1.96013)
  Week 48 (n=22) | 1.2382 (1.98754)
  Week 52 (n=22) | 1.2019 (1.71587)
  Week 56 (n=18) | 3.9651 (12.83795)
  Week 60 (n=17) | 2.6449 (8.93648)
  Week 64 (n=15) | 0.6341 (1.40213)
  Week 68 (n=11) | 0.5210 (1.49015)
  Week 72 (n=10) | 1.5263 (1.97617)
  Week 76 (n=8) | 2.0304 (2.49171)
  Week 80 (n=7) | 1.4975 (2.39680)
  Week 84 (n=7) | 11.4459 (25.92600)
  Week 88 (n=3) | 0.0704 (0.06935)
  Follow up (n=32) | 2.3169 (3.24139)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks after last actual study medication (up to 101 weeks)
Description: Analysis was performed on safety population.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 3/41
Other Adverse Events (participants affected / at risk) | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=41)
Multiple injuries (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=41)
Neutropenia (Blood and lymphatic system disorders) | 3
Pharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4

LIMITATIONS AND CAVEATS:
The study was terminated prior to the planned final on-treatment efficacy assessments due to commercial availability of tocilizumab in Russia and Poland.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.